CLINICAL TRIAL: NCT04121585
Title: Clinical Observation Study of the Hydroxylapatite-coated SL-PLUS™ Hip Shaft
Acronym: SL-PLUS HA
Status: Terminated | Type: Observational
Why Stopped: Business reasons. High subject attrition at the 10-year timepoint leading to loss of statistical power and data value. Decision finalised 24May2023.
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: D10080-3
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: HA (hydroxylapatite) coated SL-PLUS™ stem
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SL-PLUS™ hydroxylapatite coated cement free hip stem: Total Hip Arthroplasty using the SL-PLUS™ hydroxylapatite coated cement free hip stem
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — Total Hip Arthroplasty using the SL-PLUS™ hydroxylapatite coated cement free hip stem

SUMMARY:
Summary from initial protocol

Goal: Validation of the HA (hydroxylapatite) coated SL-PLUS™ stem within an observation study

Study design: prospective, multicenter, observational, non-comparative study

Study population: 240 consecutive cases (HA-coated implants), 60 cases per study site

Intervention (if applicable): Implantation of a total hip endoprosthesis Main goals/endpoints: Radiological: radiolucent lines, osteolysis, hypo- and hypertrophy of the cortex, loosening of the implant or migration; clinical: Harris Hip Score, implant-related complications, revisions; patient questionnaires HOOS and EQ-5D

Type and extent of the risks associated with the study participation as well as benefits for the patient:

All patients will benefit from the hip prostheses without exception. There are no increased risks for the patients participating in the study compared to patients who do not participate. Normal, necessary follow-up exams will be performed over the course of 10 years. These follow-up exams will then be quantitatively evaluated within the scope of the study in accordance with a standardized protocol. Accordingly, the benefit for the patients from the participation in the study is currently not yet foreseeable.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip endoprosthesis of the side affected (unilateral or bilateral)
* Patient shall be provided with a HA-coated SL-PLUS™ stem
* Patient has no general medical contraindications regarding the surgery
* Signed informed consent form for the participation in the study
* X-ray examinations are possible
* Patient is willing to participate in the post-operative follow-up program
* Age: 18-75 years

Exclusion Criteria:

* Previous failed hip joint surgery (endoprosthesis) of the side affected
* Previous infections in the joint affected; systemic infections

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 240 consecutive cases (HA-coated implants), 60 cases per study site
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-06-12 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | up to 10 years after implantation
  The Harris Hip Score (HHS) is a clinician-based outcome measure frequently used for the evaluation of patients following a total hip arthroplasty. The score considers information on pain, function and range of motion. The scale ranges from 0 - 100 whereas, a higher score indicates a favorable outcome.
WOMAC Osteoarthritis Index | up to 10 yeares after implantation
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on I off toilet, heavy domestic duties, light domestic duties
EuroQuol-5D questionnaire | up to 10 years after implantation
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal
Intra- und perioperative implant-related "Adverse Events" (AE) and complications until discharge | from surgery up to 7 days after surgery
  Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects
Postoperative AE up to 10 years after the surgery | up to 10 years after implantation
  Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects
Survival, Kaplan Meier | up to 10 years after implantation
  Hip implants in situ after 10 years of follow-up

SECONDARY OUTCOMES:
Radiographic changes | up to 10 years after implantation
  Radiographic changes defined as radiolucent lines, osteolysis, hypo- and hypertrophy of the cortex, loosening of the implant or migration.

CONTACTS AND LOCATIONS:
Overall Officials: K Zweymüller, Univ. Prof. Dr, Study Chair — Orthopädisches Krankenhaus Gersthof; Vinzenz Auersperg, Prim. Dr., Principal Investigator — Orthopädie LKH Steyr
Locations (2):
- Austria (2):
  - Orthopädie LKH Steyr, Steyr
  - Orthopädisches Krankenhaus Gersthof, Vienna

IPD SHARING:
Plan to Share IPD: No